CLINICAL TRIAL: NCT03446456
Title: The Influence of Vasopressin on Observational Learning of Placebo Analgesia
Brief Title: Vasopressin and Pain Perception in the Brain
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Luana Colloca, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HP-00076723
Record Dates: First submitted 2018-01-16; First posted 2018-02-26 (Actual); Results first posted 2021-12-16 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Acute Pain
Keywords: Magnetic Resonance Imaging; Healthy Volunteers; Arginine Vasopressin; Antidiuretic Hormone; Analgesia; Social Behavior
MeSH Terms: conditions — Acute Pain; Diabetes Insipidus; Agnosia; Social Behavior | interventions — Arginine Vasopressin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This experiment has a between-subjects design. Participants will be randomized into two groups: AVP and control. Both the experimenter and participant will be blinded to the group allocation. Participants have 50%/50% chance of being placed in either group. Participants in the AVP group will receive intranasal AVP and the participants in the control group will receive intranasal saline before the fMRI experiment. The experiment in the fMRI scanner is divided into two phases: an observational phase in which participants will observe a video of a demonstrator experiencing analgesia and a testing phase in which study participants will receive heat pain to investigate how their pain perception. During both phases there will be a placebo condition (pain with the expectation of having received a treatment) and a control condition (pain without the expectation of having received a treatment). All participants will complete both phases, including the observational and testing phase.
Who Masked: Participant, Investigator
Masking Description: Randomization will be performed/maintained by the University of Maryland Medical Center Pharmacy. Blind will only be broken in case of a potential medical emergency during the experiment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Saline (Placebo Comparator): Under direction of a research team member, participants will self-administer intranasal normal saline shortly before beginning the fMRI experiment.
  Investigators, staff, and participants were blinded to the treatment options. Each of the agents will be administrated by means of a nasal spray. Participants will be instructed by a nurse/PI to self-administer the nasal spray as follows: one spray in each nostril alternating sides, 30 seconds apart for a total of two sprays per nostril.
  Interventions: Other: Saline; Behavioral: Observational learning; Other: fMRI data aquisition
- Arginine vasopressin (Experimental): Under direction of a research team member, participants will self-administer intranasal vasopressin shortly before beginning the fMRI experiment. The of AVP will be 40IU. The quantity per unit (1 mL) of Arg8-vasopressin synthetic, manufactured by Polypeptide Group Inc. (http://www.polypeptide.com) was 0.323 mg. This amount was diluted in 0.9% sodium chloride (B. Broun Medical Inc.).
  Interventions: Drug: Arginine vasopressin; Behavioral: Observational learning; Other: fMRI data aquisition

INTERVENTIONS:
Drug: Arginine vasopressin — Intranasal vasopressin will be administered shortly before the fMRI experiment.
  Other Names: Arg8-vasopressin synthetic
  Arms: Arginine vasopressin
Other: Saline — Intranasal saline will serve as a placebo for participants in the Saline Arm
  Other Names: Placebo
  Arms: Saline
Behavioral: Observational learning — During the observational learning intervention, participants will learn the experience of analgesia in another person via a video. Participants will learn the analgesia nature of the placebo cream and the neutral nature of the control cream.
  Other Names: Social observation
Other: fMRI data aquisition — All participants from the intranasal vasopressin and intranasal saline groups will go through a fMRI data acquisition to obtain the brain structural, brain resting-states and functional MRI scans.

SUMMARY:
The feeling of pain is not just a sensory experience, but is also influenced by emotions, beliefs and expectations, making pain a highly subjective experience. This is evident in clinical practice, where the behavior of the physician and the treatment context can strongly influence the pain experience of patients. Research has shown that patients' expectation that a treatment will reduce pain influences individual perception of pain, even if the treatment has no active ingredient. The expectancy-induced analgesia emerges due to a modulation of the individual pain experience of patients by an engagement of endogenous inhibitory systems in the central nervous system.

The development of expectancy-induced analgesia can be generated in several ways. The investigators have previously demonstrated that social information and observational learning (e.g. the patient observes analgesia in another person receiving a treatment) can lead to expectancy-induced analgesia and pain reduction. However, the neural mechanisms (mechanisms in the brain) of how these expectancies are acquired and the neural mechanisms of analgesia induced by observational learning are unknown.

The investigators recently established a procedure to investigate neural mechanisms of observational learning in placebo analgesia. Here the investigators propose to investigate the influence of vasopressin, a neurotransmitter that is important for social interaction, on observational learning.

The investigators will use functional magnetic resonance imaging (fMRI), a non-invasive method, to investigate neural activity in humans. Participants will either receive vasopressin or saline with a nasal spray. During fMRI scanning, participants will then undergo an observational learning phase, where the study participants will learn the experience of analgesia in another person through a video, and a testing phase, where participants will perceive painful stimulations with the same cues as the observational phase. The comparison of the vasopressin group and the saline group will allow us to investigate how vasopressin influences behavioral effects of observational learning on pain perception as well as its effect on the neural processing of observational learning.

A better understanding of how the human brain processes observationally-induced analgesia would allow us to improve the therapeutic context of pain treatments by increasing the contextual factors which help patients cope with pain.

DETAILED DESCRIPTION:
The purpose of this research is to investigate how vasopressin (AVP) influences the neural mechanisms associated with observationally-induced analgesia. More specifically, the investigators will determine how observing another person experiencing analgesia shapes subsequent behavioral and neural responses to painful stimulations.

Aim 1: To investigate how AVP influences the neural mechanisms associated with observationally-induced analgesia.

Hypothesis 1: The investigators expect that AVP will boost activation in brain regions involved in social cognition.

The overall objective is to determine the effect of AVP on brain mechanisms associated with observationally-induced analgesia. This experiment has a between-subject study design. Participants will be randomized into an AVP group and a control group. The experimenter as well as the participant will be blinded regarding the allocation of the participant. Participants in the AVP group will receive intranasal AVP and the participants in the control group will receive intranasal saline before the fMRI experiment. Participants have 50% chance of being placed in either group. The experiment in the fMRI scanner is divided into two phases: an observational phase, in which participants will observe a video of a demonstrator experiencing analgesia, and a testing phase, in which study participants will receive heat pain to investigate how pain perception was influenced. During both phases there will be a placebo condition (pain with the expectation of having received a treatment) and a control condition (pain without the expectation of having received a treatment). All participants will complete both phases, including the observational and testing phase.

Expectancy of analgesia related to the act of receiving a treatment (e.g. a painkiller) can reduce pain perception, even if this treatment is in fact an inert substance (e.g. placebo). Expectancies about analgesic treatments can be acquired in several different ways, including direct experience of analgesia (i.e. the patient learns that after taking a specific drug, pain will decrease), verbal instructions (i.e. the doctor tells the patient that a specific drug will reduce pain) or social observation (i.e. the patient observes pain relief in another patient after this patient took a specific drug).

The direct experience of pain relief in the context of treatment cues (i.e. conditioning) reduces subsequent pain perception when the same treatment cues are present. The neural underpinnings of how treatment expectancies are acquired during conditioning have been investigated previously. These studies indicate that the prefrontal cortex is involved in learning treatment expectations in the context of conditioned analgesic effects.

However, these expectancies can also be acquired by observing others. Our group was the first to demonstrate that analgesia can be triggered by observing another person that experiences analgesia. This finding has been corroborated with additional studies by our group and other groups. In these experiments, participants acquire expectancies of analgesia not by experiencing pain relief themselves, but rather by observing another person (the demonstrator) experiencing analgesia after receiving a certain analgesic treatment (actually a sham treatment). These placebo manipulations generate expectancies which lead to placebo effects of similar sizes that those shown through direct experience via conditioning paradigms.

Even though previous research has focused on the direct experience of pain relief within a treatment context, social psychology suggests that most human behaviors are in fact modulated by sociality and learned by observing others. The investigators recently established a paradigm to investigate neural mechanisms of observational learning in placebo analgesia. The preliminary data analysis (unpublished data) suggests that while participants are observing someone else experiencing less pain due to an analgesic treatment, brain regions associated with mentalizing processes such as left and right temporoparietal junction (TPJ) and medial prefrontal cortex (mPFC) show increased activation. However, the underlying neurotransmitter systems are unknown. Here, the investigators aim to investigate how AVP modulates this network of brain regions. AVP is a likely candidate system, because recently it has been associated with placebo analgesia by my current mentor's lab, is involved in controlling a wide variety of social behaviors, and has been shown to critically modulate TPJ activity. The investigators expect that AVP will lead to increased activation of the mentalizing network during observational learning, and therefore, to increased placebo analgesia as a result of the observational learning. In order to investigate this, the investigators will perform a similar observational learning study in a group receiving intranasal AVP and a control group receiving intranasal saline.

Background: Clinical outcomes are not just related to pharmacological substances, but also to the context in which a treatment is given as well as expectancies, fears, desires and beliefs of the patient. The beneficial effects on health related outcome changes due to the treatment context and not due to specific actions of a drug are known as placebo effects. In the field of pain, the reduction of pain perception due to placebo effects is called placebo analgesia or expectancy-induced analgesia.

Previous research shows that in placebo analgesia, informational cues of the treatment context generate the expectancy of pain relief due to a treatment. These expectations can be acquired through several ways, including learning through direct experience (i.e. conditioning), verbal instruction or observation of others.

Several studies investigated the influence of direct experience of analgesia using conditioning paradigms on placebo effects. These studies show that conditioning creates more robust placebo effects than verbal suggestions alone and that the magnitude of experienced pain relief and the duration influence subsequent placebo effects.

On the neural level, placebo effects on pain perception are mediated by the descending pain modulatory system. Endogenous opioids are involved in the pain descending modulation systems, and placebo analgesia can be substantially reduced by opioid antagonists. Several studies implicate functional connectivity between the rostral anterior cingulate and the periaqueductal gray, a region critical for descending pain modulation, and placebo analgesia. Additionally, there is considerable evidence that prefrontal regions, especially the dorsolateral prefrontal cortex (DLPFC), are critically involved in placebo analgesia. The prefrontal cortex consistently shows higher activations related to the anticipation of analgesia and experience of pain relief induced by a placebo manipulation, and is involved in the acquisition of expectancies during conditioning of placebo analgesia.

Therefore the current understanding is that the prefrontal cortex maintains and updates expectancies regarding pain, and that these prefrontal regions influence the experience of pain by activating the descending pain modulatory system.

The influence of social learning on placebo analgesia has been investigated to a lesser degree. Recent research suggests that placebo analgesia can also be induced by observational learning, however, the neural neurotransmitter systems underpinning observationally-induced placebo analgesia have not yet been investigated.

Rationale: To harness the placebo effects in clinical contexts, it is important to understand how placebo effects arise and are maintained. Previous neuroscience research has primarily focused on conditioning paradigms, however human behaviors are affected by social learning. Social learning refers to learning about the environment due to information gained by observing others. Our overall hypothesis is that AVP will increase neural activation in regions related to social cognition during observational learning. Our objective is to determine the interplay of AVP and observationally-induced analgesia using an fMRI approach. fMRI is a noninvasive technique to measure changes in blood oxygenation in the brain enabling us to draw inferences about the localization and extend of neural activation associated with specific events and cues including the perception of experimental painful stimulations and modulation. The investigators designed an experiment to be performed behaviorally and with fMRI measurements in order to determine the interplay of AVP and observationally-induced analgesia.

Significance: This experiment will advance our understanding of endogenous processes associated with observationally-induced analgesia and the factors that influences pain processing. A better understanding of how treatment expectancies, formed through social observation, influence the individual experience of pain is significant in several ways. First, it will allow a better understanding of the contextual factors shaping pain and responses to treatments in clinical settings. Second, knowledge about the neural processes associated with endogenous pain relief might lead to novel developments in pain therapeutic strategies. Third, the investigators anticipate generating findings that will advance our knowledge of how cognitive processes (i.e. expectancy) are represented in the brain and how these factors influence human social behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Age ( 18-55 years old)
* English speaker (written and spoken)

Exclusion Criteria:

* Cardiovascular, neurological diseases, pulmonary abnormalities, kidney disease, liver disease, degenerative neuromuscular disease, history of cancer within past 3 years
* Any history of chronic pain disorder or currently in pain
* Severe psychiatric condition (e.g. schizophrenia, bipolar disorders, mania, autism) and /or psychiatric condition leading to treatment and/or hospitalization within the last 3 years.
* Family (first degree) history of mania, schizophrenia, or other psychoses
* Lifetime alcohol/drug dependence or alcohol/drug abuse in past 3 months
* Pregnancy or breast feeding
* Color-blindness
* Impaired, uncorrected hearing
* History of angioedema
* High blood pressure (above 140 mmHg) or symptomatic low blood pressure
* History of fainting
* Left handed
* Allergies or sensitivities to creams, lotions or food coloring
* Any non-organic implant or any non-removable metal device (e.g. pacemaker, cochlear implants, stents, surgical clips, non-removable piercings)
* Any prior eye injury or the potential of a foreign body in the eye (e.g. worked in metal fields)Persisting functional impairment due to a head trauma
* Fear of closed spaces
* Any other contraindications for MRI (e.g. large tattoos on head and neck)
* Previously participated in a "Pain Perception in the Brain" Study
* Failed drug test (testing for opiates, cocaine, methamphetamines, amphetamines and THC)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Luana Colloca, MD/PHD/MS, Principal Investigator — University of Maryland Baltimore School of Nursing
Locations (1):
- Luana Colloca, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
At this time, there is neither intent nor plan to share IPD.

REFERENCES:
- [Background] Colagiuri B, Schenk LA, Kessler MD, Dorsey SG, Colloca L. The placebo effect: From concepts to genes. Neuroscience. 2015 Oct 29;307:171-90. doi: 10.1016/j.neuroscience.2015.08.017. Epub 2015 Aug 10. PMID 26272535
- [Background] Colloca L, Benedetti F. Placebo analgesia induced by social observational learning. Pain. 2009 Jul;144(1-2):28-34. doi: 10.1016/j.pain.2009.01.033. Epub 2009 Mar 10. PMID 19278785
- [Background] Colloca L, Pine DS, Ernst M, Miller FG, Grillon C. Vasopressin Boosts Placebo Analgesic Effects in Women: A Randomized Trial. Biol Psychiatry. 2016 May 15;79(10):794-802. doi: 10.1016/j.biopsych.2015.07.019. Epub 2015 Aug 4. PMID 26321018
- [Background] Schenk LA, Sprenger C, Geuter S, Buchel C. Expectation requires treatment to boost pain relief: an fMRI study. Pain. 2014 Jan;155(1):150-157. doi: 10.1016/j.pain.2013.09.024. Epub 2013 Sep 26. PMID 24076046
- [Background] Born J, Lange T, Kern W, McGregor GP, Bickel U, Fehm HL. Sniffing neuropeptides: a transnasal approach to the human brain. Nat Neurosci. 2002 Jun;5(6):514-6. doi: 10.1038/nn849. No abstract available. PMID 11992114

RESULTS

PARTICIPANT FLOW:
Groups:
- Saline: Under direction of a research team member, participants will self-administer intranasal normal saline shortly before beginning the fMRI experiment.
  Investigators, staff, and participants were blinded to the treatment options. Each of the agents will be administrated by means of a nasal spray. Participants will be instructed by a nurse/PI to self-administer the nasal spray as follows: one spray in each nostril alternating sides, 30 seconds apart for a total of two sprays per nostril.
  Saline: Intranasal saline will serve as a placebo for participants in the Saline Arm
  Observational learning: During the observational learning intervention, participants will learn the experience of analgesia in another person via a video. Participants will learn the analgesia nature of the placebo cream and the neutral nature of the control cream.
- Arginine Vasopressin: Under direction of a research team member, participants will self-administer intranasal vasopressin shortly before beginning the fMRI experiment. The of AVP will be 40IU. The quantity per unit (1 mL) of Arg8-vasopressin synthetic, manufactured by Polypeptide Group Inc. (http://www.polypeptide.com) was 0.323 mg. This amount was diluted in 0.9% sodium chloride (B. Broun Medical Inc.).
  A random allocation sequence will be independently generated by the UM Pharmacy. The Principal investigator will call for each experiment. Participants will be first stratified for sex and then randomized to saline (0.4 mL) or vasopressin (40 IU) group, respectively.
  Arginine vasopressin: Intranasal vasopressin will be administered shortly before the fMRI experiment.
  Observational learning: During the observational learning intervention, participants will learn the experience of analgesia in another person via a video. Participants will learn the analgesia nature of the placebo cream and the neutral nature of the control cream.
Period: Overall Study
Arm/Group | Saline | Arginine Vasopressin
Started | 20 | 20
Completed | 16 | 16
Not Completed | 4 | 4
Not completed — Participant was in a previous social learning study (exclusion criteria) | 1 | 1
Not completed — Lost to Follow-up | 1 | 3
Not completed — Participant failed the toxicology test | 1 | 0
Not completed — Break down of the experimental equipment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline | Arginine Vasopressin | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.25 (7.43) | 25.44 (5.75) | 26.84 (6.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 14 | 13 | 27
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 7 | 4 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 5 | 7 | 12
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change in BOLD Singal in Supplementary Motor Area Compared to Whole Brain Average During the Painful Stimulation
Description: Blood oxygenation level dependent (BOLD) responses will allow the identification of relative activation/deactivation in the brain as a result of events (e.g. painful stimulations) that will be given during the experiment.
  Changes in the Percentage of BOLD signal are calculated as the BOLD signal in the right supplementary motor area during the 20-second heat pain divided by the whole-brain average BOLD signal during that 20-second heat pain.
Time Frame: Day 2, the average of 24 trials of painful stimulations with each stimulation lasting 20 seconds
Measure: Mean (Standard Deviation); unit: percentage of BOLD signal change
Arm/Group | Saline | Arginine Vasopressin
Number analyzed (Participants) | 16 | 16
percentage of BOLD signal change | 0.485 (0.271) | 0.482 (0.387)
Statistical Analysis 1: Comparison: Saline vs Arginine Vasopressin; Percentage of BOLD signal change was calculated as the BOLD signal in the right supplementary motor area (SMA, a typical brain area responding to pain stimulation), divided by the BOLD signal of the whole-brain average during the 24 trials of 20-second painful stimulations. The percentage of BOLD signal changes in SMA during the 20-second painful stimulations were compared between the Saline group and the Vasopressin group using an equivalence test; Test type: Equivalence — An equivalence test was conducted to compare if the vasopressin group differed from the saline group in changes of BOLD signal in the brain; p = 0.982, t-test, 2 sided — Bonferroni corrected; Mean Difference (Final Values) = 0.00264

2. Secondary Outcome: Heating Temperature
Description: On Day 1, the heating temperature was calibrated to the individual level. The heating temperature corresponding to 50 out of 100 visual analog scale pain ratings was selected as the testing temperature for day 2 (test).
Time Frame: Day 1 (calibration)
Measure: Mean (Standard Deviation); unit: celsius degree
Arm/Group | Saline | Arginine Vasopressin
Number analyzed (Participants) | 16 | 16
celsius degree | 44.16 (0.77) | 44.44 (0.83)
Statistical Analysis 1: Comparison: Saline vs Arginine Vasopressin; Test type: Equivalence — An equivalence test was conducted to compare if the vasopressin group differed from the saline group in heating temperature that was used for the testing phase; p = 0.269, ANCOVA — Bonferroni corrected; The drug group (Vasopressin vs. Saline) was set as a between-subject factor. Age and race were treated as covariates; Mean Difference (Final Values) = -0.282

3. Other Pre Specified Outcome: Implicit Association Test (IAT) Response Latency Difference
Description: The IAT is a behavioral test that examines racial biases via measuring the strength of associations between concepts (e.g., African-American, Asian, White) and evaluations (good, bad). Participants were asked to press a response key when they saw images (people) or words (good/bad) on the screen. Response latencies (RL) were measured in milliseconds using E-prime as the reaction time to press the response key. An RL difference (D) score was calculated as 1) Compute the standard deviation (SD) of RL from overall trials; 2) M1 is the mean of RL in the condition where "White" and "good" share the same response key. M2 is the mean of RL in the condition where "African-American/Asian people" and "good" share the same response key; 3) D = (M2-M1)/SD.
  The D score ranges from -2 to +2. Positive values indicate a racial preference for White people. Negative values indicate a racial preference for African-American/Black or Asian people. A value close to 0 indicates no racial preference.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: difference score
Arm/Group | Saline | Arginine Vasopressin
Number analyzed (Participants) | 16 | 16
difference score | 0.03 (0.37) | 0.07 (0.32)
Statistical Analysis 1: Comparison: Saline vs Arginine Vasopressin; Response latencies were recorded to calculate the IAT difference score (D). A difference score (D) was calculated based on the following steps: 1) Compute the standard deviation (SD) of response latencies from overall trials; 2) M1 is the mean of the response latencies in the condition where "White people" and "good" share the same response key. M2 is the mean of the latencies in the condition where "African-American/Asian people" and "good" share the same response key; 3) D = (M2-M1)/SD; Test type: Equivalence — An equivalence test was conducted to compare if the vasopressin group differed from the saline group in implicit racial biases; p = 0.378, ANCOVA; Drug group (Vasopressin vs. Saline) was set as between-subject factor. Age and race were treated as covariates; Mean Difference (Final Values) = -0.04

4. Secondary Outcome: Pain Ratings
Description: Participants will provide their pain on a Visual Analogue Scale raging from 0=no pain to 100= maximum unbearable pain. Normal value will be absence of pain.
Time Frame: Day 2 (test)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saline | Arginine Vasopressin
Number analyzed (Participants) | 16 | 16
units on a scale | 44.84 (24.49) | 47.19 (26.27)
Statistical Analysis 1: Comparison: Saline vs Arginine Vasopressin; Test type: Equivalence — An equivalence test was conducted to compare if the vasopressin group differed from the saline group in self-reported pain intensity ratings; p = 0.014, Mixed Models Analysis — Bonferroni corrected; Age, race, and heating temperature used during the testing phase were treated as covariates; Mean Difference (Final Values) = -2.35

ADVERSE EVENTS:
Time Frame: The adverse event was monitored from the time-point of drug administration to 80 minutes after the drug administration.
Arm/Group | Saline | Arginine Vasopressin
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT03446456/Prot_SAP_002.pdf
  • Informed Consent Form (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT03446456/ICF_003.pdf